CLINICAL TRIAL: NCT00017758
Title: The Effect of Efavirenz and Nelfinavir on the Pharmacokinetics of Hydroxymethylglutaryl Coenzyme A Reductase Inhibitors
Brief Title: The Effect of Efavirenz and Nelfinavir on the Blood Levels of Certain Lipid-Lowering Drugs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Purpose: Treatment
Other Study IDs: ACTG A5108; AACTG A5108
Record Dates: First submitted 2001-06-11; First posted 2001-08-31 (Estimated); Last update posted 2006-03-14 (Estimated); Status verified 2004-02

CONDITIONS: HIV Infections; HIV Seronegativity; Lipodystrophy
Keywords: Drug Interactions; Nelfinavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Pharmacokinetics; Pravastatin; efavirenz; Simvastatin; atorvastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors
MeSH Terms: conditions — HIV Infections; Lipodystrophy | interventions — Pravastatin; Simvastatin; Atorvastatin; Nelfinavir; efavirenz

INTERVENTIONS:
Drug: Pravastatin sodium
Drug: Simvastatin
Drug: Atorvastatin calcium
Drug: Nelfinavir mesylate
Drug: Efavirenz

SUMMARY:
The purpose of this study is to find out whether certain anti-HIV drugs (efavirenz [EFV] and nelfinavir [NFV]) affect the amount of certain fat-lowering drugs (atorvastatin, pravastatin, and simvastatin) in the blood.

Protease inhibitors (PIs), a type of anti-HIV drug, are known to cause increased lipids (fats) in the blood of HIV-infected patients. EFV also is known to increase blood fats. HIV-infected patients who take PIs and/or EFV may need to take fat-lowering drugs to correct this problem. So it is important to look at possible drug interactions when these drugs are taken together. This study will see if taking EFV or NFV, a protease inhibitor, affects the blood level of simvastatin, atorvastatin, or pravastatin (all fat-lowering drugs). To obtain results more quickly, the study population will be healthy HIV-negative volunteers.

DETAILED DESCRIPTION:
Abnormalities in lipid metabolism are a recognized side effect of protease inhibitor (PI) therapy in HIV-infected patients. EFV also is known to increase plasma cholesterol. In an attempt to normalize serum lipids in HIV-infected patients on PIs and/or EFV, Hydroxymethylglutaryl Coenzyme A (HMG-CoA) reductase inhibitors (also known as statins) may be prescribed. Therefore, it is important to study how PIs and EFV affect the PK of concurrently-administered statins. Many of the statins utilize the cytochrome P450 (CYP) 3A4 enzyme for metabolism. In addition, atorvastatin and simvastatin have active metabolites, generated via CYP3A4, that contribute to the drugs' lipid-lowering activity and probably to their toxicity. Pravastatin is not metabolized by CYP3A4 but is inactivated by conjugation, non-CYP3A4-induced hydroxylation, and renal excretion. NFV, the most commonly used PI, is an inhibitor of CYP3A4 and an inducer of other CYPs and conjugative pathways. EFV is a mixed CYP3A4 inhibitor and inducer. This study examines the effect of NFV on the PK of pravastatin and the effect of EFV on the PK of simvastatin, atorvastatin, and pravastatin. As EFV with pravastatin is expected to be a common drug combination during the treatment of HIV infection, it should be explored further, even though drug interactions are not expected. To expedite this study, the study population is comprised of healthy control volunteers.

Volunteers are assigned to 1 of 4 groups. Volunteers in Groups A, B, and C take a statin (simvastatin, atorvastatin, or pravastatin, respectively) on Days 0 to 3. After Day 3, the statin is stopped and EFV is begun. Volunteers take EFV until Day 14 and the statin and EFV together from Days 15 to 18. Volunteers in Group D take pravastatin on Days 0 to 3, NFV on Days 4 to 12, and pravastatin and NFV together on Days 13 to 16. Fasting lipid profiles are performed on Days 0, 4, 15, and 19 for Groups A, B, and C, and on Days 0, 3, 13, and 16 for Group D. PK sampling is performed on Days 3, 14, and 18 for Groups A, B, and C (requiring an overnight stay), and on Days 3 and 16 for Group D. Volunteers receive monetary compensation for participation in this study.

ELIGIBILITY:
Inclusion Criteria

Volunteers may be eligible for this study if they:

* Are HIV-negative.
* Are 18 to 60 years old.
* Weigh at least 50 kg (110 lbs) and are within 30 percent of their ideal body weight.
* Cannot have children (have reached menopause [change of life] for at least 24 straight months or have had a hysterectomy), if female and enrolling to Group A, B, or C.
* Have a negative pregnancy test within 14 days before study entry and within 24 hours before starting the study drugs, if female, able to have children, and enrolling to Group D.
* Agree to avoid trying to become pregnant or causing someone to become pregnant. Agree not to donate sperm or participate in other fertilization procedures. If participating in sexual activity that could lead to pregnancy, the study volunteer and/or partner must use 2 reliable methods of birth control at the same time, while taking study drugs, and for 6 weeks after stopping the drugs. Male volunteers are allowed to be sexually active without the use of birth control if they have had a successful vasectomy or are sterile.

Exclusion Criteria

Volunteers will not be eligible for this study if they:

* Have or have had heart, kidney, blood, nerve, digestive, mental, hormonal, or immune system diseases. These include high blood pressure, blocked arteries, arthritis, diabetes, stomach or intestinal problems, depression, and past use of antidepressant drugs.
* Are pregnant or breast-feeding.
* Have used experimental, prescription, or over-the-counter drugs within 14 days before study entry, except for aspirin (ASA), acetaminophen (Tylenol), diphenhydramine (Benadryl), daily multivitamins, mineral supplements, birth control pills or implants, and hormone replacement therapy for women who have reached menopause.
* Are allergic to study drugs or their ingredients.
* Abuse drugs or alcohol.
* Have a medical condition that, in the opinion of the investigator, would interfere with their participation in the study.
* Have participated in any experimental drug study within 30 days before study entry.
* Are not able to keep their usual diet during the study or are unable to write down their food intake before the study visits.
* Have an abnormal urine test result, e.g., urinary tract infection, kidney disease, or kidney stones.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56

CONTACTS AND LOCATIONS:
Overall Officials: John Gerber, Study Chair; Judith Aberg, Study Chair
Locations (10):
- United States (10):
  - Stanford Univ Med Ctr, Stanford, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Univ of Minnesota, Minneapolis, Minnesota
  - Washington Univ / St Louis Connect Care, St Louis, Missouri
  - Washington Univ School of Medicine, St Louis, Missouri
  - Univ of Rochester Medical Center, Rochester, New York
  - Univ of Cincinnati, Cincinnati, Ohio
  - Univ of Pittsburgh, Pittsburgh, Pennsylvania
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Result] Aberg JA, Rosenkranz SL, Fichtenbaum CJ, Alston BL, Brobst SW, Segal Y, Gerber JG; ACTG A5108 team. Pharmacokinetic interaction between nelfinavir and pravastatin in HIV-seronegative volunteers: ACTG Study A5108. AIDS. 2006 Mar 21;20(5):725-9. doi: 10.1097/01.aids.0000216373.53819.92. PMID 16514303